CLINICAL TRIAL: NCT06355804
Title: Lifestyle Physical Activity Intervention for Persons Newly Diagnosed With Multiple Sclerosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Robert W Motl, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY2023-1565
Record Dates: First submitted 2024-03-27; First posted 2024-04-09 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
Keywords: Physical activity; Behavior change; Behavioral intervention
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity condition (Experimental): Participants in this arm will receive a remote-delivered physical activity program for 16 weeks that includes access to electronic newsletters and regular one-on-one coaching chats (15 - 30 minutes) over Zoom with a behavioral coach after the baseline assessment. Throughout the 16-week period, The investigators will ask participants to wear a Fitbit (provided) for tracking daily physical activity.
  Interventions: Behavioral: Physical activity condition
- Waitlist condition (Other): Participants will receive access to a remote-delivered physical activity program for 16 weeks that includes access to electronic newsletters and regular one-on-one coaching chats (15-30 minutes) over Zoom with a behavioral coach after the follow-up assessment.
  Interventions: Behavioral: Waitlist condition

INTERVENTIONS:
Behavioral: Physical activity condition — Participants will receive a remote-delivered physical activity program for 16 weeks that includes access to electronic newsletters and regular chats over Zoom with a behavioral coach:
  * The newsletters provide behavioral strategies such as information on the benefits of physical activity, goal setting and monitoring, for increasing and maintaining physical activity levels.
    * Throughout the 16-week period, the investigators will ask participants to wear a Fitbit and record step count into a logbook daily for tracking physical activity.
    * The newsletter will be emailed to participants weekly throughout the program. The newsletters include knowledge, skills, and resources related to physical activity in the early stages of MS.
  * The program also involves 7 1-on-1 coaching chats with a coach to guide participants through the program and navigate challenges. These chats are conducted over Zoom and generally last about 15 - 30 minutes each. These sessions will not be recorded.
  Arms: Physical activity condition
Behavioral: Waitlist condition — Participants will receive access to a remote-delivered physical activity program for 16 weeks that includes access to electronic newsletters and regular chats over Zoom with a behavioral coach:
  * The newsletters provide information on the benefits of physical activity, goal setting and monitoring, and other behavioral strategies for increasing and maintaining physical activity levels.
    * The newsletter will be emailed to participants weekly throughout the program.
    * Content on the newsletter includes knowledge and skills related to physical activity in the early stages of MS, text of individuals with MS discussing their experiences, web links, worksheets, and brochures.
  * The program also involves 7 one-on-one video coaching chats with a behavioral coach to guide participants through the program and navigate challenges. These chats are conducted face- to-face over Zoom and generally last about 15 - 30 minutes each. The investigators do not record these sessions.
  Arms: Waitlist condition

SUMMARY:
The overall objective of the current study is to determine the efficacy of a 16-week remotely delivered lifestyle behavioral intervention compared with a control condition (i.e., waitlist control) in persons newly diagnosed with MS (disease duration ≤ 2 years).

Specific Aim 1: To evaluate the changes in self-report and device-measured physical activity after the 16-week remotely delivered physical activity behavior change intervention compared with a control condition (i.e., waitlist control) in persons who have diagnosed with MS within the past two years. The investigators hypothesize that the 16-week behavior change intervention will yield greater improvements in physical activity levels than the control condition immediately after the intervention.

Specific Aim 2: To investigate the efficacy of the 16-week, remotely delivered physical activity behavior change intervention compared with the control condition for improvements in fatigue, depression, anxiety, and QoL in persons newly diagnosed with MS. The investigators hypothesize that there will be beneficial effects on the symptoms and QoL outcomes immediately after the physical activity intervention compared with minimal changes in the control condition.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a prevalent neurological disease of the central nervous system that is the leading cause of neurological disability among young adults in the United States. This disease results in the progressive loss of walking, substantial worsening of cognition, symptoms of fatigue, as well as compromised quality of life (QoL). There is evidence that physical activity is beneficially associated with walking mobility, cognitive function, symptoms of fatigue, depression, anxiety, and pain in persons with MS. Nonetheless, this population is strikingly sedentary and physically inactive, including persons newly diagnosed with MS (diagnosed with MS for two years or less). Indeed, approximately 40% of persons with MS reported stopping physical activity after an MS diagnosis, and persons recently diagnosed with MS have not been included in physical activity intervention research. Yet, the early stage of MS represents an ideal time point for initiating physical activity for life-long benefits. There is further evidence that physical activity and exercises interventions delivered remotely can yield benefits in managing MS symptoms and comorbidities, and disability progression. To this end, the objective of this current study is to examine the efficacy of a 16-week remotely delivered behavioral intervention, compared with a control condition (i.e., waitlist control), for increasing physical activity and improving secondary outcomes in persons newly diagnosed with MS (disease duration ≤ 2 years). Participants will complete a series of assessments of physical activity, MS symptoms, and physical and cognitive function before and immediately after the 16-week program. The assessments involve the completion of a battery of questionnaires remotely over the Internet. The investigators will also ask that participants wear an accelerometer (like a pedometer) during the waking hours of the day for a 7-day period as an assessment of physical activity. The first assessments occur upon enrollment in the study (Baseline Assessment) and the second occurs right after the intervention (16- week Assessment). In this study, participants will be randomly assigned into 1 of 2 conditions: a physical activity condition (receive the intervention immediately after baseline assessment) or a waitlist condition (receive the intervention after the 16-week assessment). Participants in both conditions will receive access to an Internet delivered program for 16 weeks as well as one-on-one coaching through Zoom. The investigators will ask that participants in the physical activity condition wear a Fitbit (this is different from the accelerometer) for tracking physical activity daily during the 16- week period. The investigators will further ask that information from the Fitbit be recorded into a logbook daily.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* self-reported diagnosis of MS by a neurologist within the past 2 years
* relapse-free for the past 30 days
* ability to speak and read English as primary language
* internet and e-mail access, and willingness to complete the testing and questionnaires
* ambulatory without an assistive device (e.g., cane)
* insufficiently active (Godin Leisure-Time Exercise Questionnaire (GLTEQ) < 14)
* visual ability and literacy to read newsletter with font size 14 points
* on a disease-modifying therapy.

Exclusion Criteria:

* pregnant
* have elevated risk for undertaking strenuous or maximal exercise based on two or more affirmatives on the Physical Activity Readiness Questionnaire (PAR-Q)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Behavior | Changes in the GLTEQ scores from Baseline (pre-intervention) and after 16 weeks (post-intervention)
  Godin Leisure-Time Exercise Questionnaire (GLTEQ); scores range between 0 (min) and 119 (max), higher scores indicate greater engagement in physical activity behavior.
Physical Activity Behavior | Changes in the IPAQ scores from Baseline (pre-intervention) and after 16 weeks (post-intervention)
  International Physical Activity Questionnaire (IPAQ); scores range between 0 (min) and 107 (max), higher scores indicate greater engagement in physical activity behavior.
Physical Activity Level (Light physical activity) | Changes in time spent in LPA from Baseline (pre-intervention) and after 16 weeks (post-intervention)
  Time (minutes/day) spent in light physical activity (LPA) will be measured by a waist-worn accelerometer (ActiGraph model GT3X+); participants will wear the accelerometer on a belt around their waist during the waking hours of a 7 day period; a longer time of LPA reflects a higher level of physical activity.
Physical Activity Level (Moderate-to-vigorous physical activity) | Changes in time spent in MVPA from Baseline (pre-intervention) and after 16 weeks (post-intervention)
  Time (minutes/day) spent in moderate-to-vigorous physical activity (MVPA) will be measured by a waist-worn accelerometer (ActiGraph model GT3X+); participants will wear the accelerometer on a belt around their waist during the waking hours of a 7 day period; a longer time of MVPA reflects a higher level of physical activity.
Physical Activity Level (Daily step count) | Changes in time spent in daily step count from Baseline (pre-intervention) and after 16 weeks (post-intervention)
  Daily step count will be measured by a waist-worn accelerometer (ActiGraph model GT3X+); participants will wear the accelerometer on a belt around their waist during the waking hours of a 7 day period; a greater number of steps per day reflects a higher level of physical activity.

SECONDARY OUTCOMES:
Health-related quality of Life | Changes in SF-12 scores from Baseline (pre-intervention) and after 16 weeks (post-intervention)
  Short Form Health Status Survey (SF-12); scores range between 0 (min) and 100 (max), higher scores indicate better physical and mental aspects of quality of life.
Health-related Quality of Life | Changes in MSIS-29 scores from Baseline (pre-intervention) and after 16 weeks (post-intervention)
  Multiple Sclerosis Impact Scale (MSIS-29); scores range between 0 (min) and 100 (max), higher scores indicate greater impact of disease on daily function (i.e. worse outcomes).
Fatigue Severity | Changes in fatigue severity scores from Baseline (pre-intervention) and after 16 weeks (post-intervention)
  Fatigue Severity Scale (FSS); scores range between 1 (min) and 7 (max), higher scores reflect greater fatigue severity.
Depressive Symptoms | Changes in depressive symptoms scores from Baseline (pre-intervention) and after 16 weeks (post-intervention)
  Hospital Anxiety and Depression Scale (HADS); scores range between 0 (min) and 21 (max), higher scores reflect greater frequency of anxiety and depressive symptoms.
Anxiety | Changes in anxiety scores from Baseline (pre-intervention) and after 16 weeks (post-intervention)
  Hospital Anxiety and Depression Scale (HADS); scores range between 0 (min) and 21 (max), higher scores reflect greater frequency of anxiety and depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States